CLINICAL TRIAL: NCT04535817
Title: The Effect of Omalizumab (Xolair) on Improving Neuropsychiatric Symptoms in a Subset of ASD Patients With Atopic Disease and Elevated Total IgE Levels
Brief Title: Xolair Interventional Study in ASD Patients With Comorbid Atopy
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: We are terminating due to loss of funding because of Covid-19.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Xue-Jun Kong, Research Investigator, Beth Israel Deaconess Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020P000753
Record Dates: First submitted 2020-08-13; First posted 2020-09-02 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Autism Spectrum Disorder; Atopy
Keywords: omalizumab
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Omalizumab

STUDY DESIGN:
Intervention Model Description: Baseline testing, followed by 24-week treatment period, followed by 24-week follow-up period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment Group (Experimental): Subjects will receive subcutaneous treatment of 300mg of omalizumab during the 24-week treatment period. One injection will be administered every 4 weeks.
  Interventions: Drug: Omalizumab Injection [Xolair]

INTERVENTIONS:
Drug: Omalizumab Injection [Xolair] — 300mg via 2 subcutaneous injections every 4 weeks
  Other Names: Xolair

SUMMARY:
Following the publication of two case studies that reported behavioral benefit in ASD patients treated with omalizumab, the investigators will conduct a pilot trial to test the proof-of-concept efficacy of omalizumab in ASD patients with comorbid atopic disease. Investigators will evaluate behavioral improvement using three questionnaires. Investigators will also perform fMRI on all subjects and obtain serum samples for quantification of immunological biomarkers. If the trial is conclusive, the investigators will conduct a larger-scale, randomized-controlled trial to further understand the pathology of allergy in this subpopulation of ASD patients and the efficacy of this intervention.

DETAILED DESCRIPTION:
This clinical trial is a Phase I, single-arm, open-label study. All 20 subjects will be given the same dosage of the study drug. Following baseline testing, subjects will undergo treatment during a 24 week treatment period and will receive six subcutaneous injections total, one injection every 4 weeks. A 24-week follow-up period after the treatment period will be concluded with patient interview. Behavioral questionnaires will be administered throughout the duration of the trial. fMRI will be conducted at baseline and at the conclusion of the treatment period. Blood will be drawn for serum testing at baseline, at Week 12 during the treatment period, and at the conclusion of the treatment period. Vitals and CGI will also be assessed throughout the trial.

ELIGIBILITY:
Inclusion criteria:

* Age between 18-30 years old.
* Clinical diagnosis of ASD during childhood that is still active.
* History of atopic diseases, including asthma, atopic dermatitis, and allergic rhinitis.
* Total serum IgE level ≥ 30 IU/ml and ≤ 400 IU/ml

Exclusion criteria:

* History of omalizumab use.
* Subjects who have used oral or systemic steroid burst within 6 weeks of study enrollment. Subjects who are receiving a maintenance dose of Prednisone of 5 mg/day or less will be allowed provided the dose of Prednisone is not changed during the study.
* Subjects actively taking the antipsychotic medication, Loxapine.
* History of cancer or pre-cancer.
* Subjects with active or unstable seizure disorder.
* History or active signs of psychosis.
* Body weight > 90kg
* For subjects who meet allergic rhinitis inclusion criteria, RCAT >20
* IQ < 70
* Adaptive Behavior Composite score < 90, based on the Vineland 3rd Edition
* Lactating or pregnant females. Xolair has not been sufficiently tested for safe use in pregnant females.
* Subjects who are deemed by the study staff to be unable to cooperate with or understand the instructions that will be given during the study.
* Subjects with severe medical condition(s) that in the view of a Physician Investigator prohibits participation in the study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-01-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in Social Responsiveness Scale (SRS) Edition 2 | Baseline and Week 12
  Social communication and behavior - The scoring is based on T-score which is based on the sum of responses as follows (76 to higher - severe, 66 to 75- moderate deficiencies, 60 to 65 - mild deficiencies, 59 and below is not clinically significant for ASD).
Change from Baseline to Week 24 in Social Responsiveness Scale (SRS) Edition 2 | Baseline and Week 24
  Social communication and behavior - The scoring is based on T-score which is based on the sum of responses as follows (76 to higher - severe, 66 to 75- moderate deficiencies, 60 to 65 - mild deficiencies, 59 and below is not clinically significant for ASD).
Change from Baseline to Week 48 in Social Responsiveness Scale (SRS) Edition 2 | Baseline and Week 48
  Social communication and behavior - The scoring is based on T-score which is based on the sum of responses as follows (76 to higher - severe, 66 to 75- moderate deficiencies, 60 to 65 - mild deficiencies, 59 and below is not clinically significant for ASD).
Change from Week 24 to Week 48 in Social Responsiveness Scale (SRS) Edition 2 | Week 24 (conclusion of treatment period) and Week 48 (follow-up)
  Social communication and behavior - The scoring is based on T-score which is based on the sum of responses as follows (76 to higher - severe, 66 to 75- moderate deficiencies, 60 to 65 - mild deficiencies, 59 and below is not clinically significant for ASD).
Change from Baseline to Week 12 in Aberrant Behavior Checklist (ABC) | Baseline and Week 12
  Social behavior test - The total score is calculated based on 5 sub-scales (Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactive/Noncompliance, and Inappropriate Speech). There are 58 questions that are scored on a 0-3 scale 0 -"not at all a problem", 1- "the behavior is a problem but slight in degree", 2- "the problem is moderately serious" and 3- "the problem is severe in degree". Based on this sub-scores are calculated and added to get the total score.
Change from Baseline to Week 24 in Aberrant Behavior Checklist (ABC) | Baseline and Week 24 (conclusion of treatment period)
  Social behavior test - The total score is calculated based on 5 sub-scales (Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactive/Noncompliance, and Inappropriate Speech). There are 58 questions that are scored on a 0-3 scale 0 -"not at all a problem", 1- "the behavior is a problem but slight in degree", 2- "the problem is moderately serious" and 3- "the problem is severe in degree". Based on this sub-scores are calculated and added to get the total score.
Change from Baseline to Week 48 in Aberrant Behavior Checklist (ABC) | Baseline and Week 48 (follow-up)
  Social behavior test - The total score is calculated based on 5 sub-scales (Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactive/Noncompliance, and Inappropriate Speech). There are 58 questions that are scored on a 0-3 scale 0 -"not at all a problem", 1- "the behavior is a problem but slight in degree", 2- "the problem is moderately serious" and 3- "the problem is severe in degree". Based on this sub-scores are calculated and added to get the total score.
Change from Week 24 to Week 48 in Aberrant Behavior Checklist (ABC) | Week 24 (conclusion of treatment period) and Week 48 (follow-up)
  Social behavior test - The total score is calculated based on 5 sub-scales (Irritability, Social Withdrawal, Stereotypic Behavior, Hyperactive/Noncompliance, and Inappropriate Speech). There are 58 questions that are scored on a 0-3 scale 0 -"not at all a problem", 1- "the behavior is a problem but slight in degree", 2- "the problem is moderately serious" and 3- "the problem is severe in degree". Based on this sub-scores are calculated and added to get the total score.
Change from Baseline to Week 1 in Autism Treatment Evaluation Checklist (ATEC) | Baseline and Week 1
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.
Change from Baseline to Week 4 in Autism Treatment Evaluation Checklist (ATEC) | Baseline and Week 4
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.
Change from Baseline to Week 8 in Autism Treatment Evaluation Checklist (ATEC) | Baseline and Week 8
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.
Change from Baseline to Week 12 in Autism Treatment Evaluation Checklist (ATEC) | Baseline and Week 12
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.
Change from Baseline to Week 16 in Autism Treatment Evaluation Checklist (ATEC) | Baseline and Week 16
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.
Change from Baseline to Week 20 in Autism Treatment Evaluation Checklist (ATEC) | Baseline and Week 20
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.
Change from Baseline to Week 24 in Autism Treatment Evaluation Checklist (ATEC) | Baseline and Week 24 (conclusion of treatment period)
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.
Change from Baseline to Week 48 in Autism Treatment Evaluation Checklist (ATEC) | Baseline and Week 48 (follow-up)
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.
Change from Week 24 to Week 48 in Autism Treatment Evaluation Checklist (ATEC) | Week 24 (conclusion of treatment period) and Week 48 (follow-up)
  Social Behavior Test - The total score is calculated by adding together the scores of 4 subtests (Speech/Language Communication, Sociability, Sensory/Cognitive Awareness, and Health/Physical/Behavior). This 67 question test will provide scores for each subtest and a total score, for which a higher score indicates greater symptom severity.

SECONDARY OUTCOMES:
Inflammatory Marker Levels | Baseline, Week 12, and Week 24 (conclusion of treatment period)
  Inflammatory marker serum concentration quantification (free IgE, total IgE, interleukin 6, tumor necrosis factor alpha, tryptase).
Structural MRI | Baseline and Week 24 (conclusion of treatment period)
  The software Freesurfer will be used to calculate volume of brain regions and diffusion parameters (e.g. fractional anisotropy and mean diffusivity) from structural T1 and diffusion tensor images respectively. Paired t-test will be used to compare brain volume at baseline and post-treatment.
Functional MRI (resting state) | Baseline, and Week 24 (conclusion of treatment period)
  Correlation analysis will be used to calculate the connectivity across different brain regions. Paired t-test will be used to compare differences in activity at baseline and post-treatment.
Generalized Anxiety Disorder 7-item (GAD-7) | Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Anxiety symptom questionnaire - Scoring is based on how frequently the subject experienced 7 GAD-related symptoms in the last two weeks. Each question is rated on a 0-3 scale: 0 - "Not at all", 1 - "Several days", 2 - "More than half the days", 3 - "Nearly every day." Defined cutoffs will be used to define severity.
Epworth Sleepiness Scale (ESS) | Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Sleepiness Questionnaire - Scoring is based on how likely the subject is to doze off or fall asleep during 8 daily activities. Higher scores indicate more severe sleepiness.
Pittsburgh Sleep Quality Index (PSQI) | Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Sleep Quality Questionnaire - Scoring is based on 19 self-administered questions and 5 roommate questions. An algorithm provided with the questionnaire will be used to calculate global sleep quality score, for which a higher score indicates greater severity.
Asthma Control Test (ACT) | Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  A 5 question patient survey designed to identify patients with poorly controlled asthma based on the symptom severity over the last 4 weeks.
Rhinitis Control Assessment Test (RCAT) | Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  A 6 question patient survey designed to evaluate rhinitis symptom control based on symptom severity and frequency over the past week.
Validated Investigator Global Assessment of Atopic Dermatitis (vIGA-AD) | Baseline, Week 1, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  A clinical assessment tool used to describe severity of atopic dermatitis. The vIGA-AD includes a single scale from 0-4, in which 0 is "clear" and 4 is "severe."

OTHER OUTCOMES:
Clinical Global Impressions Scale - Improvement (CGI-I) | Baseline, Week 0, Week 4, Week 8, Week 12, Week 16, Week 20, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Psychological Clinical Assessment - Conducted by a physician, this 7-point scale characterizes changes in the subject's clinical presentation.
Clinical Global Impressions Scale - Severity (CGI-S) | Baseline, Week 0, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Psychological Clinical Assessment - Conducted by a physician, this 7-point scale defines severity of the subject's psychopathology.
Autonomic indices 1 | Baseline, Week 0, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Blood volume pulse
Autonomic indices 2 | Baseline, Week 0, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Heart Rate
Autonomic indices 3 | Baseline, Week 0, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Blood oxygen saturation
Autonomic indices 4 | Baseline, Week 0, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Carboxyhemoglobin blood saturation
Autonomic indices 5 | Baseline, Week 0, Week 4, Week 8, Week 12, Week 16, Week 20, Week 24 (conclusion of treatment period), and Week 48 (follow-up)
  Blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Jun Kong, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data with researchers not directly involved in this study and on the research team.